CLINICAL TRIAL: NCT03162003
Title: Irish Programme for Stratified Prostate Cancer Therapy
Acronym: iPROSPECT
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 14-04
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood processed to Plasma, serum and filtered for Circulating Tumour Cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patient with visceral disease and/or bone lesions (excluding patients who only have nodal disease), who have commenced or are about to commence ADT and whose disease has not shown any evidence of castration resistance.
- Cohort 2: Patient with castrate-resistant disease at time of treatment change

SUMMARY:
The purpose of the trial is to investigate new clinical tests that could predict what treatments work best for certain patients with advanced prostate cancer by identifying markers and indicators present in blood and tissue which correlate with treatment response.

DETAILED DESCRIPTION:
Prostate Cancer (PCa) is a complex disease and not all patients respond to every treatment available.

This study aims to investigate new clinical tests based on simple and routine blood tests to allow men with PCa and their doctors to choose the correct treatment for their metastatic PCa.

In this way, only men likely to respond to the specific treatment will be chosen, sparing unnecessary or prolonged treatment for those who will not respond and allowing them to avail of alternative therapies likely to have more benefit. This is termed personalised therapy.

The study will perform research on biological elements present in the blood including deoxyribonucleic acids (DNA), ribonucleic acid (RNA), protein and circulating tumour cells (CTCs) which are cancer cells that have spread beyond the prostate gland and can be found floating in the blood. Clinical data will be correlated to research findings to form conclusions on personalised therapy.

Additional optional sub studies include; magnetic resonance imaging (MRI) with a biopsy of another tumour in a different site of their body such as bone, lung or liver (metastatic biopsy), metastatic biopsy only and biopsies of the fluid of solid part of the bone. These optional components provide more detailed information on prostate cancer and how men are responding to treatment. The research results from these optional sub studies will be correlated with the research analysis from the blood samples and clinical data and will help to make treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 4 mPCa as confirmed by CT/MRI or by bone scan
2. Patient with visceral disease and/or bone lesions (excluding patients who only have nodal disease), who have commenced or are about to commence ADT and whose disease has not shown any evidence of castration resistance (cohort 1) Or Patient with castrate-resistant disease at time of treatment change (cohort 2)
3. Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 28 days prior to recruitment
4. Life expectancy of at least 6 months
5. Ability to give written informed consent obtained before any study-related procedures
6. Age ≥ 18 years and male

Exclusion Criteria:

1. Diagnosis of or treatment for another systemic malignancy within 2 years before study entry.*
2. Any evidence of residual disease from a previously diagnosed malignancy. *Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with castrate sensitive (cohort 1) or castrate resistant (cohort 2) metastatic prostate cancer.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Androgen Deprivation Therapy (ADT) alone and combined. | 10 years
  Identification of predictive biomarkers for ADT treatment or ADT combined treatment response in metastatic prostate cancer
Biomarkers to treatment response | 10 years
  Identification of predictive biomarker(s) for treatment response in metastatic castrate resistant prostate cancer

SECONDARY OUTCOMES:
Circulating Tumour Cells (CTC's) | 10 years
  Analysis of the biology of CTCs from metastatic prostate cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Ray McDermott, Principal Investigator — SVUH, AMNCH
Locations (9):
- Ireland (9):
  - Cork University Hospital, Wilton road, Cork
  - Adelaide and Meath Hospital incorporating the National Children's Hospital (AMNCH), Tallaght, Dublin
  - Beacon Hospital, Sandyford, Dublin
  - Beaumont Hospital, Beaumont, Dublin
  - Mater Misericordiae University Hospital & Mater Private Hospital, Dublin
  - St James's Hospital, James's street, Dublin
  - St Vincent's University Hospital, Elm Park, Dublin
  - Sligo University Hospital, The Mall, Sligo
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: No